CLINICAL TRIAL: NCT06704919
Title: Assess Clinical and Radiographic Outcomes of Conduit Cages and Fibergraft in Cervical and Lumbar Procedures
Brief Title: Conduit Cages and Fibergraft BG Putty
Status: Recruiting | Type: Observational
Sponsor: Nitin Agarwal (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Sponsor-Investigator, Nitin Agarwal, Associate Professor, Neurosurgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY24040009
Record Dates: First submitted 2024-10-28; First posted 2024-11-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Degenerative Disc Disease; Herniated Disc
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Use of conduit cages and fibergraft BG Putty — Patients who require spine surgery under standard of care and meet the inclusion and exclusion criteria identified, will be recruited from clinic. Consent for participation in study will be signed at the same time as consent for surgery. All PROMs and scans will be done as standard of care and data will be obtained through chart review for this study.

SUMMARY:
The Conduit cages are intended to restore the intervertebral height and to facilitate the intervertebral body fusion in the cervical and lumbar spine in skeletally mature patients with degenerative disc disease and instabilities at one or more levels of the spine. The Fibergraft Bioactive Glass (BG) is engineered to mimic the body's natural bone healing process. While previous studies have described the use of conduit cages in interbody fixation procedures, these studies did not specifically study the clinical and radiographic outcomes of patients who have received these implants in addition to Fibergraft. We aim to recruit patients with degenerative disc disease, and instabilities at one to multilevel contiguous levels between C2-T1 and 1-2 contiguous levels between L2-S1 of the spine with accompanying radicular symptoms, ruptured or herniated discs, and pseudarthrosis and spondylodesis. We will then follow these patients for a duration of two years to report their clinical and radiographic outcomes to determine fusion, complication rate, and revision surgeries if any.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Have a radiograph-based diagnosis of degenerative disc disease, ruptured or herniated discs,
3. Pathology of the cervical or lumbar spine.
4. Pathology to be between C2-T1 in the cervical group.
5. Pathology to be between L2-S1 in the lumbar group.
6. Patients with 1-2 contiguous levels in both ACDF and Lumbar groups.
7. Patients receiving the surgery/devices as standard of care prescribed by the treating physician.

Exclusion Criteria:

1. Patients < 18 years
2. BMI > 40 kg/m2 to be excluded
3. Patients with a bone density (DEXA) score of <2.0 to be excluded
4. 3 or more levels for ACDF or Lumbar interbody to be excluded
5. Patients with previous pseudoarthrosis or failed spondylodesis to be excluded
6. Current smokers and patients who quit smoking within 6 weeks prior to presentation will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with spinal conditions mentioned in inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Fusion | 2 years (At baseline, postoperatively at 6 weeks, 3 months, 6 months, 12 months, and 24 months)
  We will assess fusion with regular x-rays and CT scans at 1 and 2-year postoperatively.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 2 years (At baseline, postoperatively at 6 weeks, 3 months, 6 months, 12 months, and 24 months)
  We will have patients fill out validated tools for PROs to assess how the patient is doing postoperatively
Oswestry Disability Index | 2 years (At baseline, postoperatively at 6 weeks, 3 months, 6 months, 12 months, and 24 months)
  We will have patients fill out validated tools for PROs to assess how the patient is doing
SF-12 | 2 years (At baseline, postoperatively at 6 weeks, 3 months, 6 months, 12 months, and 24 months)
  We will have patients fill out validated tools for PROs to assess how the patient is doing
Neck Disability Index | 2 years (At baseline, postoperatively at 6 weeks, 3 months, 6 months, 12 months, and 24 months)
  We will have patients fill out validated tools for PROs to assess how the patient is doing

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Agarwal, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No